CLINICAL TRIAL: NCT05788549
Title: The Effect of Progressive Relaxation Techniques on Disease Activity, Anxiety, Sleep, and Quality of Life in Individuals With Ulcerative Colitis
Brief Title: Assessment of the Effectiveness of Progressive Relaxation Techniques in Individuals With Ulcerative Colitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Yağmur ARTAN, Research Assistant, PhD student, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-1T/50
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Progressive relaxation techniques; Quality of Life; Sleep Quality; Anxiety; Disease activity
MeSH Terms: conditions — Colitis, Ulcerative; Sleep Initiation and Maintenance Disorders; Anxiety Disorders | interventions — Autogenic Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Progressive Relaxation Group (Experimental): The Individual Identification Form, Partial Mayo Score, State-Trait Anxiety Inventory, Pittsburgh Sleep Quality Index, and IBD-QOL were filled out in person during the first meeting. The first application was done face to face with the researcher. Individuals were asked to perform subsequent applications at home.Educational booklet describing the progressive relaxation exercises with pictures was given to individuals, and a video prepared by the researcher was uploaded to their mobile phones. Individuals were asked to practice progressive relaxation exercises every day, at least once a day, in a quiet and peaceful environment for 30-minute sessions. The researcher sent reminder SMS messages to individuals twice a week for eight weeks to encourage regular practice of the progressive relaxation exercises. Four and eight weeks after the first meeting, forms were transferred to an online environment and sent to individuals via WhatsApp Messenger as a link to be completed
  Interventions: Behavioral: Progressive Muscle Relaxation
- Relaxative Music Group (Placebo Comparator): The Individual Identification Form, Partial Mayo Score, State-Trait Anxiety Inventory, Pittsburgh Sleep Quality Index, and IBD-QOL were filled out in person during the first meeting. Individuals were asked to perform subsequent applications at home.Individuals were provided with a relaxing music file prepared by the researcher and were asked to listen to it at least once a day for 30 minutes in a quiet and calm environment. The researcher also sent reminder SMS messages twice a week for eight weeks to remind individuals. Four and eight weeks after the first meeting, forms were transferred to an online environment and sent to individuals via WhatsApp Messenger as a link to be completed to listen to the relaxing music regularly. At 4 and 8 weeks after the first meeting, the researcher transferred the forms to an online environment via Google Forms and asked individuals to fill them out by accessing the link sent to them via WhatsApp Messenger
  Interventions: Behavioral: Relaxative Music
- Control Group (No Intervention): The Individual Identification Form, Partial Mayo Score, State-Trait Anxiety Inventory, Pittsburgh Sleep Quality Index, and IBD-QOL were filled out in person during the first meeting.The members of this group have not undergone any intervention and continued their routine maintenance, treatment, and follow-up.At 4 and 8 weeks after the first meeting, the researcher transferred the forms to an online environment via Google Forms and asked individuals to fill them out by accessing the link sent to them via WhatsApp Messenger

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation — The Individual Identification Form, Partial Mayo Score, State-Trait Anxiety Inventory, Pittsburgh Sleep Quality Index, and IBD-QOL were filled out in person during the first meeting. The first application was done face to face with the researcher. Individuals were asked to perform subsequent applications at home.Educational booklet describing the progressive relaxation exercises with pictures was given to individuals, and a video prepared by the researcher was uploaded to their mobile phones. Individuals were asked to practice progressive relaxation exercises every day, at least once a day, in a quiet and peaceful environment for 30-minute sessions. The researcher sent reminder SMS messages to individuals twice a week for eight weeks to encourage regular practice of the progressive relaxation exercises. Four and eight weeks after the first meeting, forms were transferred to an online environment and sent to individuals via WhatsApp Messenger as a link to be completed
  Arms: Progressive Relaxation Group
Behavioral: Relaxative Music — The Individual Identification Form, Partial Mayo Score, State-Trait Anxiety Inventory, Pittsburgh Sleep Quality Index, and IBD-QOL were filled out in person during the first meeting. Individuals were asked to perform subsequent applications at home.Individuals were provided with a relaxing music file prepared by the researcher and were asked to listen to it at least once a day for 30 minutes in a quiet and calm environment. The researcher also sent reminder SMS messages twice a week for eight weeks to remind individuals. Four and eight weeks after the first meeting, forms were transferred to an online environment and sent to individuals via WhatsApp Messenger as a link to be completed to listen to the relaxing music regularly. At 4 and 8 weeks after the first meeting, the researcher transferred the forms to an online environment via Google Forms and asked individuals to fill them out by accessing the link sent to them via WhatsApp Messenger
  Arms: Relaxative Music Group

SUMMARY:
Ulcerative colitis is a chronic disease that follows a course of remission and flare-ups. Especially during flare-ups, the worsening of symptoms negatively affects all aspects of the individual's life and decreases their quality of life. Individuals sometimes have difficulty accessing healthcare facilities. In addition, every hospital admission causes an additional burden on healthcare institutions and the individual, both physically and financially. Therefore, it is of great importance to support and develop self-management behaviors for individuals to control their symptoms.

Progressive relaxation techniques are a relaxation method based on the principle of voluntary contraction and relaxation of muscle groups in our body. It has been reported that progressive relaxation techniques, which are applied in many chronic diseases and procedures, improve symptoms and disease parameters reported by individuals, especially pain, anxiety, and stress.

When the literature in the world and Turkey is examined, no study applying progressive relaxation techniques to ulcerative colitis patients has been encountered. It is known that especially stress and anxiety affect the number and severity of flare-ups in ulcerative colitis patients. It is thought that this study will contribute to the self-management behaviors of ulcerative colitis patients in the rare diseases group for the Turkish population and fill the gap in the literature.

DETAILED DESCRIPTION:
The purpose of the research is to investigate the effect of progressive relaxation techniques on disease clinical activity, anxiety, sleep, and quality of life in individuals with ulcerative colitis.

We assigned 56 patients who met the inclusion criteria to the progressive relaxation group, the relaxing music group, and the control group using stratified randomization. The intervention (progressive relaxation) group was provided with a booklet and shown a video about progressive relaxation techniques.For the placebo (relaxing music) group, music from MusiCure, which consists of sounds of nature, was played. Reminder SMS messages were sent twice a week to the intervention and placebo groups. No intervention was administered to the control group.Forms were filled out again by individuals in the intervention, placebo, and control groups at the fourth and eighth week.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with UC at least six months ago
* Having been taking medication for at least three months
* Willingness to participate in the study
* Being 18 years of age or older
* Having been in remission for at least 3 months according to the partial Mayo score (Mayo score <2)
* Being able to use a computer, internet, and mobile phone
* Residing in Izmir or surrounding cities
* Being cooperative and able to communicate

Exclusion Criteria:

* Patients with advanced comorbid conditions such as cancer, diabetes, and chronic obstructive pulmonary disease have been excluded from the study due to the potential for more pronounced effects on symptoms and disease activity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
"State and Trait Anxiety Inventory" scores | A total of two months of progressive relaxation techniques practice for each patient
  Decreased "State and Trait Anxiety Inventory"scores of intervention group in follow-up measurements after progressive relaxation techniques intervention
"IBD-QOL" scores | A total of two months of progressive relaxation techniques practice for each patient
  Increased "IBD-QOL" scores of intervention group in follow-up measurements after progressive relaxation techniques intervention
"The Pittsburgh Sleep Quality Index" scores | A total of two months of progressive relaxation techniques practice for each patient
  Increased "The Pittsburgh Sleep Quality Index" scores of intervention group in follow-up measurements after progressive relaxation techniques intervention
" Disease Activity" scores | A total of two months of progressive relaxation techniques practice for each patient
  Increased "Disease Activity" scores of intervention group in follow-up measurements after progressive relaxation techniques intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin YILDIRIM, Prof., Study Chair — Ege University Faculty of Nursing
Locations (1):
- Ege University Faculty of Nursing, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391